CLINICAL TRIAL: NCT05729594
Title: Systemic Pharmacokinetic Study of T4032 (Unpreserved Bimatoprost 0.01%) Eye Gel Versus Lumigan® 0.01% Eye Drops in 40 Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LT4032-101
Record Dates: First submitted 2023-01-25; First posted 2023-02-15 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T4032 (Experimental)
  Interventions: Drug: Bimatoprost Ophthalmic
- Lumigan (Active Comparator)
  Interventions: Drug: Bimatoprost Ophthalmic

INTERVENTIONS:
Drug: Bimatoprost Ophthalmic — eyedrops

SUMMARY:
This study is being performed to compare the systemic pharmacokinetic profiles of T4032 and Lumigan 0.01% given that T4032 has a different formulation (in terms of excipients) from the reference product.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study
* Participants with no ocular symptoms

Exclusion Criteria:

* History of ocular trauma, infection, or inflammation within the last 3 months
* Presence of an ocular pathology such as blepharitis, conjunctivitis, uveitis, or any other ocular infection or inflammation
* IOP <10 mmHg or >21 mmHg

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of bimatoprost and bimatoprost free acid at each timepoint (in ng/mL) | at 2 timepoint : Baseline and week 2
Ocular and systemic adverse events | up to week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Newark, New Jersey, United States